CLINICAL TRIAL: NCT01081132
Title: A Phase 3, Double-blind, Randomized, Multi-center, Placebo Controlled, Dose-optimization Study Evaluating the Safety, Efficacy, and Tolerability of Once Daily Dosing With Extended-release Guanfacine Hydrochloride in Adolescents Aged 13-17 Years Diagnosed With Attention-deficit/Hyperactivity Disorder (ADHD)
Brief Title: Dose-optimization in Adolescents Aged 13-17 Diagnosed With Attention-deficit/Hyperactivity Disorder (ADHD) Using Extended-release Guanfacine HCl
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPD503-312; 2011-002221-21 (EudraCT Number)
Record Dates: First submitted 2010-03-03; First posted 2010-03-05 (Estimated); Results first posted 2014-05-23 (Estimated); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Attention-Deficit/Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Guanfacine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Extended-release Guanfacine HCl (Experimental)
  Interventions: Drug: Extended-release Guanfacine Hydrochloride
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Extended-release Guanfacine Hydrochloride — The test product will be provided as 1, 2, 3, and 4mg tablets. Subjects will be administered a once-daily dose between 1-7mg/day depending on weight.
  Other Names: Intuniv
  Arms: Extended-release Guanfacine HCl
Other: Placebo — Matching placebo will be provided as 1,2,3, and 4mg tablets. Subjects will be administered a once-daily dose of placebo between 1-7mg/day depending on weight.
  Arms: Placebo

SUMMARY:
To assess the efficacy of optimized Extended-release Guanfacine Hydrochloride compared with placebo in the treatment of adolescents aged 13-17 years with a diagnosis of ADHD as measured by the ADHD-RS-IV

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 13-17 years at the time of consent/assent (screening only).
2. Subject's parent or legally authorized representative (LAR) must provide signature of informed consent, and there must be documentation of assent by the subject indicating that the subject is aware of the investigational nature of the study and the required procedures and restrictions in accordance with the International Conference on Harmonisation (ICH) Good Clinical Practice (GCP) Guidance E6 (1996) and applicable regulations before completing any study-related procedures at screening.
3. Subject meets Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition-Text Revision (DSM-IV-TR) criteria for a primary diagnosis of ADHD, combined subtype, or hyperactive/impulsive subtype, based on a detailed psychiatric evaluation using the Kiddie Schedule for Affective Disorders and Schizophrenia - Present and Lifetime version (K SADS PL) at screening (re-confirm if baseline visit is >35 days from screening).
4. Subject has a minimum ADHD-RS-IV total score of 32 at baseline.
5. Subject has a minimum CGI-S score of 4 at baseline.
6. Subject is functioning at an age-appropriate level intellectually, as deemed by the Investigator.
7. Subject and parent/LAR understand, are able, willing and likely to fully comply with the study procedures and restrictions defined in this protocol.
8. Subject is able to swallow intact tablets.
9. All females must have a negative serum beta human Chorionic Gonadotropin (hCG) pregnancy test at screening and a negative urine pregnancy test at baseline. Female subjects must abstain from sexual activity that could result in pregnancy or agree to use acceptable methods of contraception.
10. Subject has a supine and standing blood pressure (BP) measurement within the 95th percentile for age, gender, and height.

Exclusion Criteria:

1. Subject has a current, controlled (requiring a prohibited medication or behavioral modification program) or uncontrolled, comorbid psychiatric diagnosis [except Oppositional Defiant Disorder (ODD), but including all anxiety disorders (except simple phobias)], all major depressive disorders (dysthymia allowed unless medication required), and any severe comorbid Axis II disorders or severe Axis I disorders such as post traumatic stress disorder, bipolar illness, psychosis, pervasive developmental disorder, obsessive-compulsive disorder, substance abuse disorder, or other symptomatic manifestations that, in the opinion of the Investigator, contraindicate SPD503 treatment or confound efficacy or safety assessments.
2. Subject has any condition or illness including clinically significant abnormal screening laboratory values which, in the opinion of the Investigator, represents an inappropriate risk to the subject and/or could confound the interpretation of the study.
3. Subject has a known history or presence of structural cardiac abnormalities, serious heart rhythm abnormalities, syncope, cardiac conduction problems (e.g., clinically significant heart block), exercise-related cardiac events including syncope and pre-syncope, or clinically significant bradycardia.
4. Subject has any abnormal or clinically significant ECG findings as judged by the Investigator with consideration of the central ECG interpretation.
5. Subject with orthostatic hypotension or a known history of controlled or uncontrolled hypertension.
6. Current use of any prohibited medication, including herbal supplements that affect blood pressure, heart rate, have central nervous system (CNS) effects, or affect cognitive performance, such as sedating antihistamines and decongestant sympathomimetics (inhaled bronchodilators are permitted) or a history of chronic use of sedating medications (i.e., antihistamines) at baseline.
7. Subject has a history of alcohol or other substance abuse or dependence, as defined by DSM IV-TR (with the exceptions of nicotine) within the last six months.
8. Subject has taken another investigational product within 30 days prior to baseline.
9. Subject is significantly overweight based on Center for Disease Control and Prevention Body Mass Index (BMI)-for-age gender specific charts at screening. Significantly overweight is defined as a BMI >95th percentile for this study.
10. Body weight of less than 34.0kg or greater than 91.0kg at screening.
11. Subject has a known or suspected allergy, hypersensitivity, or clinically significant intolerance to guanfacine hydrochloride or any components found in SPD503.
12. Clinically important abnormality on urine drug and/or alcohol screen (excluding the subject's current ADHD stimulant if applicable).
13. Subject is female and is pregnant or currently lactating.
14. Subject failed screening or was previously enrolled in this study.
15. Subject who is currently considered a suicide risk, has previously made a suicide attempt, or has a prior history of, or is currently demonstrating suicidal ideation.
16. History of failure to respond to an adequate trial (consisting of an appropriate dose and adequate duration of therapy), in the opinion of the Investigator, of an α2-agonist for the treatment of ADHD.
17. Subject has a history of a seizure disorder (other than a single childhood febrile seizure occurring before the age of 3 years) or a history of a tic disorder (including Tourette's syndrome).

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 314 (Actual)
Dates: Start 2011-09-19 (Actual); Primary Completion 2013-05-16 (Actual); Study Completion 2013-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (54):
- United States (54):
  - Harmonex Neuroscience Research, Dothan, Alabama
  - Clinical Study Centers, LLC, Little Rock, Arkansas
  - Peninsula Research Associates, Rolling Hills Estates, California
  - Psychiatric Centers at San Diego (PCSD-Feighner Research Institute), San Diego, California
  - Encompass Clinical Research, Spring Valley, California
  - Elite Clinical Trials, Inc., Wildomar, California
  - IMMUNO International Research Centers, Centennial, Colorado
  - Coastal Connecticut Research LLC, New London, Connecticut
  - Florida Clinical Research Center, LLC, Bradenton, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - Amedica Research Institute, Inc., Hialeah, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - George M. Joseph, MD, PA, Jacksonville Beach, Florida
  - Morteza Nadjafi, MD, FAPA, Orlando, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Miami Research Associates, South Miami, Florida
  - Janus Center for Psychiatric Research, West Palm Beach, Florida
  - Northwest Behavioral Research Center, Roswell, Georgia
  - Institute for Behavioral Medicine, Smyrna, Georgia
  - Capstone Clinical Research, Libertyville, Illinois
  - AMR-Baber Research Inc., Naperville, Illinois
  - Goldpoint Clinical Research, LLC, Indianapolis, Indiana
  - Clinco, Inc., Terre Haute, Indiana
  - Psychiatric Associates, Overland Park, Kansas
  - Four Rivers Clinical Research, Inc., Paducah, Kentucky
  - Rochester Center for Behavioral Medicine, Rochester Hills, Michigan
  - Clinical Neurophysiology Services, PC, Sterling Heights, Michigan
  - Comprehensive Psychiatric Associates, Gladstone, Missouri
  - St Charles Psychiatric Associates - Midwest Research Group, Saint Charles, Missouri
  - Center for Psychiatry and Behavioral Medicine, Inc., Las Vegas, Nevada
  - Albuquerque Neuroscience Inc., Albuquerque, New Mexico
  - Finger Lakes Clinical Research, Rochester, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Triangle Neuropsychiatry, Durham, North Carolina
  - NorthCoast Clinical Trials, Beachwood, Ohio
  - The Ohio State University, Columbus, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Tulsa Clinical Research, LLC, Tulsa, Oklahoma
  - OCCI, Inc., Portland, Oregon
  - Oregon Center for Clinical Investigations, Inc., Salem, Oregon
  - CRI Worldwide, Philadelphia, Pennsylvania
  - University Services Sleep Diagnostic and Treatment Centers, West Chester, Pennsylvania
  - Rainbow Research, Barnwell, South Carolina
  - The Jackson Clinic, Jackson, Tennessee
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Research Strategies of Memphis, LLC, Memphis, Tennessee
  - FutureSearch Trials, Austin, Texas
  - InSite Clinical Research, DeSoto, Texas
  - R/D Clinical Research, Inc., Lake Jackson, Texas
  - Westex Clinical Investigations, Lubbock, Texas
  - Neuroscience, Inc., Herndon, Virginia
  - Alliance Research Group, Richmond, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - East Side Therapeutic Resource, Kirkland, Washington

REFERENCES:
- [Derived] Wilens TE, Robertson B, Sikirica V, Harper L, Young JL, Bloomfield R, Lyne A, Rynkowski G, Cutler AJ. A Randomized, Placebo-Controlled Trial of Guanfacine Extended Release in Adolescents With Attention-Deficit/Hyperactivity Disorder. J Am Acad Child Adolesc Psychiatry. 2015 Nov;54(11):916-25.e2. doi: 10.1016/j.jaac.2015.08.016. Epub 2015 Sep 15. PMID 26506582

RESULTS

PARTICIPANT FLOW:
Groups:
- PLACEBO: Orally administered a once-daily dose
- SPD503: Orally administered a once-daily optimal dose between 0.05 mg/kg/day - 0.12 mg/kg/day (up to 7 mg/day depending on weight).
Period: Overall Study
Arm/Group | PLACEBO | SPD503
Started | 157 | 157
Completed | 102 | 105
Not Completed | 55 | 52
Not completed — Lack of Efficacy | 25 | 9
Not completed — Withdrawal by Subject | 13 | 16
Not completed — Lost to Follow-up | 4 | 11
Not completed — Adverse Event | 3 | 9
Not completed — Non Compliance | 4 | 2
Not completed — Lack Of Compliance | 0 | 1
Not completed — Missed Visits | 1 | 1
Not completed — Stopped Taking Meds | 2 | 0
Not completed — Patient Did Not Complete Wk14 and 15 | 0 | 1
Not completed — Declined Taper Phase | 0 | 1
Not completed — Protocol Violation | 3 | 1

BASELINE CHARACTERISTICS:
Population: Used Safety Population which is defined as all randomized subjects who took at least 1 dose of investigational product. Two subjects did not take investigational product, therefore n = 312.
Groups:
- Total: Total of all reporting groups
Arm/Group | PLACEBO | SPD503 | Total
Number analyzed (Participants) | 155 | 157 | 312
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.6 (1.44) | 14.5 (1.35) | 14.5 (1.39)
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 155 | 157 | 312
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 54 | 110
  Male | 99 | 103 | 202
Region of Enrollment [Count of Participants; unit: Participants] — All randomized subjects (n = 314) who received at least 1 dose of investigational product during this study.
  Participants
    UNITED STATES | 155 | 157 | 312

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Attention Deficit Hyperactivity Disorder Rating Scale-fourth Edition (ADHD-RS-IV) Total Score at Week 13
Description: The ADHD-RS-IV consists of 18 items scored on a 4-point scale ranging from 0 (no symptoms) to 3 (severe symptoms) with total score ranging from 0 to 54.
Time Frame: Baseline through week 13
Population: The Full Analysis Set consisted of all randomized subjects who took at least 1 dose of investigational product. A mixed model repeated measures (MMRM) was used to analyze the observed change from the Baseline Visit scores at all post-baseline, pre-taper, on-treatment visits.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | PLACEBO | SPD503
Number analyzed (Participants) | 106 | 109
units on a scale | -18.527 (1.0841) | -24.552 (1.0625)
Statistical Analysis 1: Comparison: PLACEBO vs SPD503; Test type: Superiority or Other; p < 0.001, Mixed Models Repeated Measures Analysis; Mean Difference (Final Values) = -6.026, 95% CI 2-sided [-8.865 to -3.187]

2. Secondary Outcome: Percent of Subjects With an Assessment of Normal/Borderline Mentally Ill on Clinical Global Impression-Severity of Illness (CGI-S) Scale at the Last On-Treatment Assessment
Description: CGI-S assesses the severity of the subject's condition on a 7-point scale: 1 (normal, not at all ill), 2 (borderline mentally ill), 3 (mildly ill), 4 (moderately ill), 5 (markedly ill), 6 (severely ill), 7 (among the most extremely ill)
Time Frame: Baseline through week 13
Population: Full Analysis Set consisted of all randomized subjects who took at least 1 dose of investigational product.
Measure: Number; unit: percentage of subjects
Arm/Group | PLACEBO | SPD503
Number analyzed (Participants) | 155 | 154
percentage of subjects | 36.1 | 50.6
Statistical Analysis 1: Comparison: PLACEBO vs SPD503; Test type: Superiority or Other; p = 0.010, Cochran-Mantel-Haenszel

3. Secondary Outcome: Change From Baseline in the Weiss Functional Impairment Rating Scale - Parent Report (WFIRS-P) Learning and School Domain Scores at Week 13
Description: The WFIRS-P is a 50-item scale with each item scored from 0 (never/not at all) to 3 (very often/very much). The Learning and School Domain consists of 10-items. Mean scores range from 0 to 3. Higher scores indicate greater functional impairment.
Time Frame: Baseline and week 13
Population: Full Analysis Set consisted of all randomized subjects who took at least 1 dose of investigational product.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | PLACEBO | SPD503
Number analyzed (Participants) | 101 | 97
units on a scale | -0.457 (0.058) | -0.572 (0.058)
Statistical Analysis 1: Comparison: PLACEBO vs SPD503; Test type: Superiority or Other; p = 0.104, Mixed Models Repeated Measures Analysis; Mean Difference (Final Values) = -0.115, 95% CI 2-sided [-0.254 to 0.024]

4. Secondary Outcome: Change From Baseline in the WFIRS-P Family Domain Score at Week 13
Description: The WFIRS-P is a 50-item scale with each item scored from 0 (never/not at all) to 3 (very often/very much). The Family Domain consists of 10-items. Mean scores range from 0 to 3. Higher scores indicate greater functional impairment.
Time Frame: Baseline and week 13
Population: Full Analysis Set consisted of all randomized subjects who took at least 1 dose of investigational product.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | PLACEBO | SPD503
Number analyzed (Participants) | 101 | 105
units on a scale | -0.314 (0.055) | -0.371 (0.054)
Statistical Analysis 1: Comparison: PLACEBO vs SPD503; Test type: Superiority or Other; p = 0.408, Mixed Models Repeated Measures Analysis; Mean Difference (Final Values) = -0.057, 95% CI 2-sided [-0.192 to 0.078]

5. Secondary Outcome: Change From Baseline in the WFIRS-P Behavior in School Domain Score at Week 13
Description: The WFIRS-P is a 50-item scale with each item scored from 0 (never/not at all) to 3 (very often/very much). Mean scores range from 0 to 3. Higher scores indicate greater functional impairment.
Time Frame: Baseline and week 13
Population: Full Analysis Set consisted of all randomized subjects who took at least 1 dose of investigational product.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | PLACEBO | SPD503
Number analyzed (Participants) | 101 | 97
units on a scale | -0.376 (0.051) | -0.459 (0.050)
Statistical Analysis 1: Comparison: PLACEBO vs SPD503; Test type: Superiority or Other; p = 0.176, Mixed Models Repeated Measures Analysis; Mean Difference (Final Values) = -0.083, 95% CI 2-sided [-0.203 to 0.037]

6. Secondary Outcome: Change From Baseline in the WFIRS-P Global Domain Score at Week 13
Description: as for outcome 5
Time Frame: Baseline and week 13
Population: Full Analysis Set consisted of all randomized subjects who took at least 1 dose of investigational product.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | PLACEBO | SPD503
Number analyzed (Participants) | 105 | 108
units on a scale | -0.296 (0.036) | -0.347 (0.035)
Statistical Analysis 1: Comparison: PLACEBO vs SPD503; Test type: Superiority or Other; p = 0.253, Mixed Models Repeated Measures Analysis; Mean Difference (Final Values) = -0.050, 95% CI 2-sided [-0.136 to -0.036]

7. Secondary Outcome: Change From Baseline in the WFIRS-P Risk Domain Score at Week 13
Description: The WFIRS-P is a 50-item scale with each item scored from 0 (never/not at all) to 3 (very often/very much). The Risk Domain consists of 10-items. Mean scores range from 0 to 3. Higher scores indicate greater functional impairment.
Time Frame: Baseline and week 13
Population: Full Analysis Set consisted of all randomized subjects who took at least 1 dose of investigational product.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | PLACEBO | SPD503
Number analyzed (Participants) | 105 | 107
units on a scale | -0.194 (0.027) | -0.191 (0.026)
Statistical Analysis 1: Comparison: PLACEBO vs SPD503; Test type: Superiority or Other; p = 0.912, Mixed Models Repeated Measures Analysis; Mean Difference (Final Values) = 0.004, 95% CI 2-sided [-0.061 to 0.068]

8. Secondary Outcome: Change From Baseline in the WFIRS-P Social Domain Score at Week 13
Description: The WFIRS-P is a 50-item scale with each item scored from 0 (never/not at all) to 3 (very often/very much). The Social Domain consists of 7-items. Mean scores range from 0 to 3. Higher scores indicate greater functional impairment.
Time Frame: Baseline and week 13
Population: Full Analysis Set consisted of all randomized subjects who took at least 1 dose of investigational product.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | PLACEBO | SPD503
Number analyzed (Participants) | 105 | 108
units on a scale | -0.234 (0.046) | -0.263 (0.045)
Statistical Analysis 1: Comparison: PLACEBO vs SPD503; Test type: Superiority or Other; p = 0.606, Mixed Models Repeated Measures Analysis; Mean Difference (Final Values) = -0.029, 95% CI 2-sided [-0.139 to 0.081]

9. Secondary Outcome: Change From Baseline in the WFIRS-P Child Self-Concept Domain Score at Week 13
Description: The WFIRS-P is a 50-item scale with each item scored from 0 (never/not at all) to 3 (very often/very much). The Child Self-Concept Domain consists of 3-items. Mean scores range from 0 to 3. Higher scores indicate greater functional impairment.
Time Frame: Baseline and week 13
Population: Full Analysis Set consisted of all randomized subjects who took at least 1 dose of investigational product.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | PLACEBO | SPD503
Number analyzed (Participants) | 104 | 106
units on a scale | -0.376 (0.067) | -0.275 (0.066)
Statistical Analysis 1: Comparison: PLACEBO vs SPD503; Test type: Superiority or Other; p = 0.228, Mixed Models Repeated Measures Analysis; Mean Difference (Final Values) = 0.102, 95% CI 2-sided [-0.064 to 0.268]

10. Secondary Outcome: Change From Baseline in the WFIRS-P Life Skills Domain Score at Week 13
Description: The WFIRS-P is a 50-item scale with each item scored from 0 (never/not at all) to 3 (very often/very much). The Life Skills Domain consists of 10-items. Mean scores range from 0 to 3. Higher scores indicate greater functional impairment.
Time Frame: Baseline and week 13
Population: Full Analysis Set consisted of all randomized subjects who took at least 1 dose of investigational product.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | PLACEBO | SPD503
Number analyzed (Participants) | 105 | 107
units on a scale | -0.328 (0.046) | -0.375 (0.045)
Statistical Analysis 1: Comparison: PLACEBO vs SPD503; Test type: Superiority or Other; p = 0.410, Mixed Models Repeated Measures Analysis; Mean Difference (Final Values) = -0.047, 95% CI 2-sided [-0.159 to 0.065]

11. Secondary Outcome: Change From Baseline in the WFIRS-P Academic Performance Domain Score at Week 13
Description: as for outcome 5
Time Frame: Baseline and week 13
Population: Full Analysis Set consisted of all randomized subjects who took at least 1 dose of investigational product.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | PLACEBO | SPD503
Number analyzed (Participants) | 104 | 96
units on a scale | -0.632 (0.096) | -0.841 (0.096)
Statistical Analysis 1: Comparison: PLACEBO vs SPD503; Test type: Superiority or Other; p = 0.082, Mixed Models Repeated Measures Analysis; Mean Difference (Final Values) = -0.208, 95% CI 2-sided [-0.443 to 0.026]

12. Secondary Outcome: Percent of Subjects With Improvement on Clinical Global Impression-Improvement (CGI-I) Scores at the Last On-Treatment Assessment
Description: Clinical Global Impression-Improvement (CGI-I) consists of a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved) or 2 (much improved) on the scale.
Time Frame: weeks 1 through 13
Population: Full Analysis Set consisted of all randomized subjects who took at least 1 dose of investigational product.
Measure: Number; unit: percentage of subjects
Arm/Group | PLACEBO | SPD503
Number analyzed (Participants) | 155 | 154
percentage of subjects | 45.8 | 67.5
Statistical Analysis 1: Comparison: PLACEBO vs SPD503; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

13. Secondary Outcome: Changes From Baseline in Behavior Rating Inventory of Executive Function (BRIEF) Scores at Week 13
Description: Behavior Rating Inventory of Executive Function (BRIEF) is a questionnaire composed of three indices: Global Executive Composite, Behavioral Regulation Index, and Metacognition Index. Items are rated 1 (never), 2 (sometimes), and 3 (often). The Global Executive Composite consists of 72 items with scoring ranging from 72 to 216. The Behavioral Regulation Index score is the total of 28 items and ranges from 28 to 84. The Metacognition Index score is the total of 44 items and ranges from 44 to 132. Lower scores reflect better functioning.
Time Frame: Baseline and week 13
Population: Full Analysis Set consisted of all randomized subjects who took at least 1 dose of investigational product.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | PLACEBO | SPD503
Number analyzed (Participants) | 82 | 88
units on a scale
  Global Executive Composite | -10.6 (1.23) | -12.9 (1.19)
  Behavioral Regulation Index | -11.5 (1.29) | -12.4 (1.25)
  Metacognition Index | -8.9 (1.18) | -11.6 (1.14)
Statistical Analysis 1: Comparison: PLACEBO vs SPD503; Global Executive Composite; Test type: Superiority or Other; p = 0.134, Mixed Models Repeated Measures Analysis; Mean Difference (Final Values) = -2.3, 95% CI 2-sided [-5.3 to 0.7]
Statistical Analysis 2: Comparison: PLACEBO vs SPD503; Behavioral Regulation Index; Test type: Superiority or Other; p = 0.579, Mixed Models Repeated Measures Analysis; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-4.0 to 2.3]
Statistical Analysis 3: Comparison: PLACEBO vs SPD503; Metacognition Index; Test type: Superiority or Other; p = 0.072, Mixed Models Repeated Measures Analysis; Mean Difference (Final Values) = -2.7, 95% CI 2-sided [-5.6 to 0.2]

14. Secondary Outcome: Change From Baseline in Pediatric Daytime Sleepiness Scale (PDSS) Total Score at Week 13
Description: The Pediatric Daytime Sleepiness Scale (PDSS) is an 8 item questionnaire scored on a scale from 0 (never) to 4 (always/very often). Total scores range from 0 to 32, with increasing score reflecting greater sleepiness.
Time Frame: Baseline through week 13
Population: Safety Population consisted of all randomized subjects who took at least 1 dose of investigational product.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | PLACEBO | SPD503
Number analyzed (Participants) | 105 | 108
units on a scale | -3.7 (0.52) | -4.2 (0.51)
Statistical Analysis 1: Comparison: PLACEBO vs SPD503; Test type: Superiority or Other; p = 0.465, Mixed Models Repeated Measures Analysis; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.8 to 0.8]

15. Secondary Outcome: Change From Baseline in Brief Psychiatric Rating Scale for Children (BPRS-C) Total Score at Last On-Treatment Assessment
Description: The BPRS-C characterizes childhood behavioral and emotional symptomatology. A total of 21 items are rated on a scale from 0 (not present) to 6 (extremely severe) with a total score ranging from 0 to 126. A decrease in score indicates a reduction in psychopathology.
Time Frame: Baseline and week 13
Population: Safety Population consisted of all randomized subjects who took at least 1 dose of investigational product.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PLACEBO | SPD503
Number analyzed (Participants) | 151 | 151
units on a scale | -7.0 (9.85) | -9.1 (8.11)

16. Secondary Outcome: Structure Side-Effect Questionnaire (SSEQ)
Description: The Structured Side-effect Questionnaire is a simple checklist of 17 side effects. The subject indicates whether a side effect has occurred since the last visit by marking 'yes' or 'no' on the checklist for each of the events listed.
Time Frame: Through week 16
Population: Safety Population consisted of all randomized subjects who took at least 1 dose of investigational product.
Measure: Number; unit: participants
Arm/Group | PLACEBO | SPD503
Number analyzed (Participants) | 155 | 157
participants
  Nausea | 33 | 37
  Vomiting | 17 | 18
  Diarrhea | 24 | 29
  Abdominal pain | 28 | 30
  Decreased appetite | 42 | 48
  Increased appetite | 47 | 42
  Headache | 53 | 76
  Dizziness | 31 | 49
  Fatigue | 43 | 65
  Nervousness/anxiety | 23 | 30
  Insomnia | 25 | 28
  Somnolence | 26 | 41
  Depression | 17 | 14
  Itching | 9 | 11
  Rash | 7 | 6
  Missed menses | 1 | 4

17. Secondary Outcome: Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS is a semi-structured interview that captures the occurence, severity, and frequency of suicide-related thoughts and behaviors during the assessment period. The interview includes definitions and suggested questions to solicit the type of information needed to determine if a suicide-related thought or behaviour occurred. The assessment is done by the nature of the responses, not by a numbered scale.
Time Frame: Through week 16
Population: Safety Population consisted of all randomized subjects who took at least 1 dose of investigational product.
Measure: Number; unit: participants
Arm/Group | PLACEBO | SPD503
Number analyzed (Participants) | 155 | 154
participants
  Suicidal ideation | 4 | 5
  Suicidal behavior | 0 | 0

ADVERSE EVENTS:
Description: Safety Population defined as all randomized subjects who took at least 1 dose of investigational product. Two subjects did not take investigational product, therefore n = 312 (Placebo = 155, SPD503 = 157).
Arm/Group | PLACEBO | SPD503
Serious Adverse Events (participants affected / at risk) | 2/155 | 4/157
Other Adverse Events (participants affected / at risk) | 120/155 | 147/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLACEBO (N=155) | SPD503 (N=157)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Homicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Withdrawal hypertension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLACEBO (N=155) | SPD503 (N=157)
Abdominal pain (Gastrointestinal disorders) | 6 (7) | 9 (10)
Abdominal pain upper (Gastrointestinal disorders) | 7 (7) | 10 (11)
Diarrhoea (Gastrointestinal disorders) | 13 (15) | 12 (17)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 12 (12)
Nausea (Gastrointestinal disorders) | 21 (22) | 19 (22)
Vomiting (Gastrointestinal disorders) | 10 (12) | 9 (9)
Fatigue (General disorders) | 19 (21) | 35 (41)
Irritability (General disorders) | 6 (6) | 11 (13)
Nasopharyngitis (Infections and infestations) | 9 (9) | 18 (20)
Upper respiratory tract infection (Infections and infestations) | 12 (14) | 14 (15)
Decreased appetite (Metabolism and nutrition disorders) | 21 (24) | 23 (27)
Increased appetite (Metabolism and nutrition disorders) | 13 (15) | 14 (15)
Dizziness (Nervous system disorders) | 16 (17) | 25 (32)
Dizziness postural (Nervous system disorders) | 3 (3) | 8 (8)
Headache (Nervous system disorders) | 28 (43) | 42 (64)
Sedation (Nervous system disorders) | 3 (3) | 18 (21)
Somnolence (Nervous system disorders) | 33 (39) | 69 (102)
Insomnia (Psychiatric disorders) | 6 (7) | 14 (16)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 3 (4)

LIMITATIONS AND CAVEATS:
For the secondary outcomes, the p-values are not controlled for multiplicity, therefore they should be considered as descriptive not inferential.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.